CLINICAL TRIAL: NCT01166204
Title: Concurrent and Non-concurrent Chemo-radiotherapy or Radiotherapy Alone With IMRT for Stage I-III Non-small Cell Lung Cancer to an Individualised MLD
Brief Title: Concurrent and Non-concurrent Chemo-radiotherapy or Radiotherapy Alone With Intensity-modulated Radiotherapy (IMRT) for Non Small Cell Lung Cancer (NSCLC) to an Individualised Mean Lung Dose (MLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRONC CONCURR MLD/BRONC MLD
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Stage I-III Non-small Cell Lung Cancer
Keywords: Radiotherapy; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group (Experimental)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy

SUMMARY:
Our group has shown that increasing the radiation dose to pre-specified normal tissue dose constraints could lead to increased TCP with the same NTCP in patients with non-concurrent and concurrent chemo-radiation. Here, the investigators want to investigate its efficacy in a prospective study in patients with stage I-III NSCLC, who are selected for high-dose radiotherapy with or without chemotherapy, but treated with IMRT. The latter technique has become standard, but the patterns of recurrence and the possibility for dose-escalation in an individualised setting have never been investigated properly.

DETAILED DESCRIPTION:
Eligible patients (see below) will receive radiotherapy to the primary tumor and the initially involved mediastinal lymph nodes to an MLD (Mean Lung Dose) of 20 +/-1Gy, irrespective of lung function.

Other dose-constraints: spinal cord max: 54Gy, brachial plexus (Dmax):66Gy

In concurrence with chemotherapy, radiotherapy will be delivered as follows:

* First three weeks/30 fractions: twice-daily fractions of 1.5Gy, with 8h to 10h as interfraction interval, 5 days per week. Total dose: 45Gy/30 fractions
* Thereafter: once daily fractions of 2.0Gy, 5 days per week until the target dose has been reached.

In sequential or radiotherapy alone schedules, twice-daily 1.8Gy with an interfraction interval of at least 8h will be delivered.

The radiation doses will be specified according to ICRU 50. Lung density corrections will be applied, as well as all standard QA procedures. Technical requirements are the same as in standard practice at MAASTRO clinic

Chemotherapy schedules allowed:

1. 1-2 cycles induction chemotherapy: any third generation schedule is allowed. The type will be registered.
2. Concurrent part: (day 1 = first day of radiotherapy)

   * cisplatin - vinorelbine
   * cisplatin - docetaxel
   * cisplatin - etoposide
   * cisplatin - pemetrexed in non-squamous histologies Q 3 weeks; 3 cycles

When the calculated creatinin clearance is less than 60ml/min, cisplatin may be substituted for carboplatin

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven NSCLC
* IUCC stage I-III, or solitary metastases (<6), which are amendable for radical local treatment.
* Performance status 0-2
* IMRT technique

Exclusion Criteria:

* Not NSCLC or mixed NSCLC and other histologies (e.g. small cell carcinoma)
* Stage IV, except for solitary (<6) metastases
* Performance status 3 or more
* No IMRT technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2.3 and 5 years

SECONDARY OUTCOMES:
Progression-free survival | 2.3 and 5 years
Dyspnea (CTCAE 4.0) | 2.3 and 5 years
Dysphagia (CTCAE 4.0) | 2.3 and 5 years
Patterns of recurrence | 2.3 and 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands